CLINICAL TRIAL: NCT05509959
Title: Women SHINE: Addressing Syndemics and HIV Among Women Through Tech-Based Peer Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jamila K. Stockman, Professor and Vice Chief, Global Public Health Section, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 210509; R01MH125785 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-08-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HIV/AIDS
Keywords: HIV Care Continuum; Psychoeducation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Placebo Comparator): Women assigned to the control arm (n=180) will receive one 60-minute group session facilitated by the licensed clinical therapist (LCT) on self-care and well-being as it relates to HIV, interpersonal violence, trauma, adverse mental health, and substance use. During this session, women will be provided with resources to HIV care, interpersonal violence, trauma, mental health, and substance use, through a static website created for Women SHINE. The content will include: 1) names and locations of clinics and organizations, services provided, and contact information; 2) links to support websites and hotlines and 3) testimonials from WLHA.
  Interventions: Behavioral: Control
- Women SHINE (Experimental): Women SHINE consists of a four-month intervention that includes video-based one-on-one peer navigation and 7 weekly psycho-education support group sessions co-facilitated by a licensed clinical therapist (LCT) and peer navigator (PN). 180 women will be enrolled in the Women SHINE intervention and will remain in their assigned psycho-education support group sessions with the same members over the course of the intervention.
  Interventions: Behavioral: Women SHINE

INTERVENTIONS:
Behavioral: Women SHINE — Minimum of nine weekly one-on-one peer navigation sessions and 7 weekly psychoeducation support group sessions.
  Arms: Women SHINE
Behavioral: Control — Single group session and access to website
  Arms: Control Arm

SUMMARY:
A two-arm RCT will be conducted to test the efficacy of Women SHINE, a web-based trauma-informed peer navigation-social support intervention (Figure 2). A total of 360 women living with HIV/AIDS (WLHA) with a history of adulthood interpersonal violence who have been prescribed ART but are non-adherent (< 90% ART adherent in the last 4 weeks) will be enrolled in the study. WLHA will be randomized (1:1) into one of the following conditions: 1) Women SHINE intervention arm (n=180) or 2) Control arm (n=180). The Women SHINE intervention arm will receive a four-month intervention including peer navigator (PN) one-on-one sessions, phone/text-based check-ins, 7 psychoeducation weekly support group sessions (120 mins.) co-facilitated by a licensed therapist and PN, and access to a static website with resources for HIV care, interpersonal violence, trauma, mental health, and substance use. The control arm will receive one group session (60 mins.) on self-care and well-being and access to the aforementioned website with resources. Women will complete a video-based survey and mailed hair sample self-collection at baseline, 4-, 8-, and 12-months post-randomization, to evaluate improvements in ART adherence (Aim 1), emotion regulation, and PTSD symptoms (Aim 2). Investigators will examine the mediating effect of individual (retention in HIV care, coping self-efficacy, social support, ancillary support services use) and socio-structural (stigma, medical mistrust) mechanisms of change on the efficacy of Women SHINE (Aim 3).

DETAILED DESCRIPTION:
In the US, women living with HIV/AIDS (WLHA) are less likely to be adherent to antiretroviral therapy (ART) and virally suppressed compared to men living with HIV/AIDS. Concurrently, WLHA experience high rates of interpersonal violence - physical, sexual, and/or psychological abuse in childhood or adulthood - which often results in trauma (e.g., post-traumatic stress disorder [PTSD]) and other adverse mental health, further contributing to ART non-adherence. Additionally, the confluence of syndemic or co-occurring adverse mental health, substance use, and socio-structural factors (e.g., HIV stigma, medical mistrust) further contribute to poor HIV outcomes. Social support through peer navigation and networks has been shown to counter these effects and improve HIV outcomes among WLHA. Likewise, psychoeducation addressing affective distress to improve mood and emotion management and relationship skills has been shown to reduce PTSD and depression. However, limited resources at HIV service agencies combined with socio-structural barriers (e.g., social isolation, lack of transportation) impede the potential effectiveness of in-person peer navigation. A scalable and sustainable solution is the use of technology in the form of web-based video interaction. Building on these promising pilot findings, investigators propose to conduct a randomized clinical trial of Women SHINE (new name) to improve ART adherence among WLHA affected by interpersonal violence in California, Arizona, and Nevada. Participants will be randomized to either: a) the intervention arm (n=180) where they will receive a 4-month program comprised of video-based peer navigation support via one-on-one sessions, 7 psychoeducation weekly support group sessions, and access to a static Women SHINE website with statewide resources for HIV care, interpersonal violence, trauma, mental health, and substance use; or b) the control arm (n=180) where they will receive a single group session on self-care and well-being, with access to the static Women SHINE website. Women will complete video-based survey assessments and mailed hair sample self-collection at baseline, 4-, 8-, and 12-months post-randomization. Compared to the control arm, investigators will determine if Women SHINE is associated with improvements in ART adherence (Aim 1) and PTSD symptoms and emotion regulation (Aim 2). Investigators will also examine individual (e.g., self-efficacy for coping, social support networks) and socio-structural (e.g., HIV stigma, medical mistrust) mechanisms of change in the efficacy of Women SHINE (Aim 3). If efficacious, investigators will conduct subsequent research to determine effective and feasible methods for intervention implementation nationwide to improve HIV outcomes among WLHA.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender female
* Diagnosis of HIV by a physician, healthcare provider, or community health worker
* Aged 18 years or older
* Speaking and reading English or Spanish
* Adulthood experiences of interpersonal violence
* Currently prescribed ART
* Self-report of <90% past-month ART adherence
* Not currently participating in another adherence intervention
* Access to an internet browser

Exclusion Criteria:

* Unwillingness to participate in the intervention
* Transgender female
* No diagnosis of HIV by a physician, healthcare provider, or community health worker
* Aged less than 18 years
* Not speaking and reading English or Spanish
* Not currently prescribed ART
* Self-report of >= 90% past-month ART adherence
* Currently participating in another adherence intervention
* No access to an internet browser
* Cognitive impairment limiting the ability to provide informed consent
* Experiencing only childhood experiences of interpersonal violence
* Inability to safely participate in the study based on secondary screener

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in ART Adherence | 4-, 8-, and 12-month post-randomization
  Adherence to ART regime measured by tenofovir (TFV), emtricitabine (FTC) concentration in hair samples
Change in ART Adherence | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of ART adherence (3 items)
Change in PTSD Symptoms | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of PTSD (9 items;PCL-5)
Change in Emotion Regulation | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of emotion regulation (16 items; DERS-16)
Change in Individual and Socio-Structural Mechanisms of Change | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of retention in HIV care
Change in Individual and Socio-Structural Mechanisms of Change | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of coping self-efficacy (26 items; CSE)
Change in Individual and Socio-Structural Mechanisms of Change | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of social support (8 items; mMOS-SS)
Change in Individual and Socio-Structural Mechanisms of Change | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of ancillary support utilization (26 items; adapted from CDC medical monitoring project), HIV stigma (30 items), and medical mistrust (12 items; GBMMS)
Change in Individual and Socio-Structural Mechanisms of Change | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of HIV stigma (30 items), and medical mistrust (12 items; GBMMS)
Change in Individual and Socio-Structural Mechanisms of Change | 4-, 8-, and 12-month post-randomization
  Validated self-report measure of medical mistrust (12 items; GBMMS)

CONTACTS AND LOCATIONS:
Overall Officials: Jamila K Stockman, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- The Regents of the Univ. of Calif., U.C. San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No